CLINICAL TRIAL: NCT00187928
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Efficacy and Safety of Adjunctive Topiramate in the Treatment of Obsessive-Compulsive Disorder
Brief Title: Study to Determine the Efficacy and Safety of Adjunctive Topiramate in the Treatment of Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ortho-McNeil Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CAPSS-217
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Obsessions; Compulsions; Adjunctive treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Obsessive Behavior; Compulsive Behavior | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to determine if a drug called topiramate is safe and effective as an add-on therapy in the treatment of Obsessive-Compulsive Disorder (OCD). Topiramate is an investigational drug for OCD, which means it has not been approved by the U.S. Food and Drug Administration (FDA). Topiramate has been approved as an add-on therapy for adults and children with partial onset seizures or generalized tonic-clonic seizures, and for patients 2 years of age and older with a severe form of epilepsy called Lennox-Gastaut Syndrome.

Up to 96 subjects will be enrolled in this study. This study consists of three phases: Washout/Screening Phase, Double-Blind Phase, and Taper Phase. The total expected length of your participation in the study is approximately four months.

DETAILED DESCRIPTION:
This is a multicenter, outpatient, randomized, double-blind, placebo-controlled, parallel-group, study designed to evaluate the safety and efficacy of adjunctive topiramate in treating subjects with OCD. The study consists of a washout/screening phase, a double-blind treatment phase of 12 weeks, a taper period of approximately 7 days. Upon successful completion of the washout/screening phase subjects will be randomized into 1 of 2 treatment groups: topiramate up to 400 mg/day or placebo. A placebo control will be used to establish the frequency and magnitude of changed in clinical endpoints that may occur in the absence of active treatment.

During the double-blind phase, subjects will be seen weekly for the first two weeks and then every other week for the remainder of the double-blind phase. Study medication will be titrated over the 8-week titration period up to 400mg/day or the subject's maximum tolerated dose. After the titration period, the dose will remain stable for the maintenance period during which visits will occur every 14 days. At the completion of the maintenance period, subjects will taper their study medication over the next 7 days.

This study will be conducted in up to 96 subjects with a diagnosis of OCD with an onset at least 1 year prior to screening supported by the SCID-I. Forty-eight subjects will be assigned to topiramate and 48 will be assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have onset of OCD at least 1 year prior to Screening (Visit 1) and must be supported by the Structured Clinical Interview for DSM-IV for Axis I Disorders (SCID-I).
2. Subjects must be taking a clinically effective dose of a Selective Serotonin Reuptake Inhibitor (SSRI) (i.e., Paroxetine, Sertraline, Fluvoxamine, Fluoxetine, Citalopram) for at least 12 weeks. Subjects must be on their current dose for at least 6 weeks and must maintain their current dose throughout the study.
3. Subjects must have stable OCD symptoms and must have a minimum severity of greater than or equal to 18 on Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) or a minimum score of greater than or equal to 10 on questions one through five if the subject has obsessions without compulsions at Visit 2 (Baseline).
4. Subjects must be between 18 and 65 years of age, inclusive.
5. Subjects can be male or female and must be in generally good health as confirmed by medical history, baseline psychiatric history and physical examination, including vital signs. Baseline laboratory values must be within normal limits, or considered clinically insignificant by the investigator.
6. Subjects must have observed the designated washout periods for prohibited medications outlined under the Concomitant Therapy section of this protocol.
7. Subjects must have a negative urine drug screening (phencyclidine, cocaine, amphetamines, tetrahydrocannabinol, and opiates) at Visit 1.
8. If female, the subject must:

   * be postmenopausal for at least one year, or
   * have had a hysterectomy or bilateral tubal ligation with resection or otherwise be incapable of pregnancy, or
   * have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, spousal/partner sterility or
   * be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence.
9. Female subjects of childbearing potential must have negative urine pregnancy test up to 7 days prior to Visit 2 (Day 1).
10. Subjects must be able to take oral medication, adhere to medication regimens and be willing to return for regular visits.
11. Subjects must be able to read and comprehend written instructions and willing to complete all scales and inventories required by this protocol.
12. After full explanation of the study, subjects must demonstrate their willingness to participate by signing an informed consent form.

Exclusion Criteria:

1. Subjects whose primary OCD symptom is hoarding. Hoarding is the most disabling and most distressing or clinically significant symptom.
2. Subjects who have a current or recent (within 6 months of the start of study medication)DSM-IV-TR diagnosis of substance dependence or abuse (with the exception of nicotine or caffeine dependence).
3. Subjects with a current or lifetime DSM-IV-TR diagnosis of bipolar disorders, or other psychotic disorder as defined by DSM-IV-TR.
4. Subjects with a history of personality disorder (e.g., schizotypal or borderline) considered by the investigator to likely interfere with assessment or compliance with treatment.
5. Subjects who are currently receiving behavioral therapy under medical supervision.
6. Subjects with prior non-response to topiramate in the opinion of the investigator for the treatment of OCD following an adequate trial.
7. Subjects who have previously been treated with topiramate and discontinued treatment due to an adverse event or subjects with a history of allergic hypersensitivity reaction to topiramate.
8. Subjects with clinically unstable disease: cardiovascular, renal, hepatic, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease that could interfere with the diagnosis, treatment, or assessment of OCD.
9. Subjects with a history of seizures.
10. Subjects with a history of nephrolithiasis.
11. Subjects with an estimated creatinine clearance of less than or equal to 60 mL/min.
12. Subjects who have SGOT and/or SGPT levels greater than 2 times the upper limit of the normal range at Visit 1.
13. Subjects who have active liver disease.
14. Subjects with progressive or degenerative neurologic disorders (e.g., multiple sclerosis).
15. Subjects known to have clinically significant medical conditions, including but not limited to:

    * symptomatic coronary artery or peripheral vascular disease
    * malignancy or history of malignancy within the past 5 years, except basal cell carcinoma;
    * any disease or condition that compromises the function of those body systems that could result in altered absorption, excess accumulation or impaired metabolism or excretion of topiramate;
    * subjects who are considered to represent a significant risk of suicidal or violent behavior in the judgement of the Investigator
16. Female subjects who are pregnant or lactating.
17. Subjects who have not observed the designated washout periods for any of the prohibited medications outlined in the Concurrent Therapy section of the protocol.
18. Subjects who in the opinion of the investigator should not be enrolled in the study because of the Precautions, Warnings or Contraindications sections of the topiramate package insert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2003-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert E Ward, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Science Center, Gainesville, Florida, United States